CLINICAL TRIAL: NCT05783336
Title: An Inter-disciplinary Approach to Understanding and Intervening on Contextual Factors That Shape HIV-risk for Young Women and Men in South Africa: Phase 2 - the Feasibility, Acceptability and Potential Effect Size of a Pilot Randomised Controlled Trial
Brief Title: Stepping Stones and Creating Futures Plus Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Medical Research Council, South Africa (Other); University College, London (Other)
Responsible Party: Principal Investigator, Andrew Gibbs, Senior Lecturer, University of Exeter
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC023-10/2022
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Intimate Partner Violence; Poverty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSCF+ (Experimental): Stepping Stones and Creating Futures Plus (SSCF+). Small group intervention, comprising approximately 15 sessions (each session ~3 hours), addressing gender, livelihoods, mental health.
  Interventions: Behavioral: Stepping Stones and Creating Futures Plus (SSCF+)
- Control (No Intervention): No intervention control (wait-list)

INTERVENTIONS:
Behavioral: Stepping Stones and Creating Futures Plus (SSCF+) — Group-based intervention delivered to small friendship networks, by a facilitator.
  Arms: SSCF+

SUMMARY:
The goal of this randomised controlled clinical trial is to test the Stepping Stones and Creating Futures Plus (SSCF+) intervention, in young (18-25 years) people living in urban informal settlements in Durban and rural communities in KwaZulu-Natal, South Africa. The main questions it aims to answer are:

* Is the intervention acceptable and feasible
* What is the potential effect size on key outcomes of intimate partner violence

Participants will be randomised (1:1) to compare SSCF+ and a control arm to see if there are differences between the two on intimate partner violence.

DETAILED DESCRIPTION:
Intimate partner violence is very common in South Africa, particularly urban informal settlements. We have co-developed an intervention, called Stepping Stones and Creating Futures Plus (SSCF+), which will be evaluated in women and men aged 18-25 years living in KwaZulu-Natal, South Africa.

This is a pilot randomised controlled trial and as such there is focus on understanding whether the intervention is acceptable (to participants), feasible to deliver, and the potential effect sizes we may see in a full trial.

ELIGIBILITY:
Inclusion Criteria:

* Normally resident in the community where recruiting
* Aged 18-30 years old
* Not in formal employment, or full-time education
* Able to communicate in the main languages of the study (English, isiXhosa or isiZulu)
* Able to provide informed consent

Exclusion Criteria:

* Only in the community temporarily
* Unable to provide informed consent
* Under 18 years of age, or over 31 years old at point of recruitment
* Unable to communicate in main study languages

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Physical Intimate Partner Violence | 6 months
  Past 6 month experience (women) and perpetration (men) of physical IPV as assessed using WHO measure of IPV (5 items, binary)
Sexual Intimate Partner Violence | 6 months
  Past 6 month experience (women) and perpetration (men) of sexual IPV as assessed using WHO measure of IPV (3 items)
Severe Intimate partner violence | 6 months
  Past 6 month experience (women) and perpetration (men) of severe IPV as assessed using WHO IPV scale (8 items, coded into a binary)

SECONDARY OUTCOMES:
Depressive symptoms | 6 months
  Mean score of depressive symptoms as assessed by the Center for Epidemiology Studies Depression Scale (CESD) comprising 20 items
Post-traumatic-stress symptoms | 6 months
  Post traumatic stress symptoms experienced in past week (mean) as assessed through the Harvard Trauma Questionnaire (16 items)
Emotional Dysregulation | 6 months
  Assessed via the Difficulties in Emotional Regulation Scale (DERS) short form, 16 items. Mean score.
Earnings | 6 months
  Self-reported past month earnings (South African Rand)
Savings | 6 months
  Self-report past month savings (South African Rand)
Hunger | 6 months
  Past month food insecurity assessed through the 3 items of the Household Food Insecurity Access Scale (HFIAS)
Livelihood Activities | 6 months
  Frequency of livelihood strengthening activities in the past 3 months, assessed through seven items
Work stress | 6 months
  Experience of stress because of lack of work and money assessed through 4 items
Work shame | 6 months
  Experience of shame because of lack of work and money assessed through 4 items
Capabilities | 6 months
  Experience of capabilities assessed through 5 items of a modified ICECAP scale

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jewkes, Principal Investigator — Medical Research Council, South Africa; Andrew Gibbs, Principal Investigator — University of Exeter; Jenevieve Mannell, Principal Investigator — University College, London
Locations (1):
- South African Medical Research Council, Durban, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared within 12 months of study completion on University of Exeter and South African Medical Research Council data repository.
Supporting Information: Study Protocol
Time Frame: 12 months from completion of study
Access Criteria: Freely available

REFERENCES:
- [Derived] Gibbs A, Washington L, Mkhwanazi S, Chirwa E, Khaula S, Shai NJ, Willan S, Batura N, Burgess R, Mnandi N, Simelane N, Jewkes R, Mannell J. Stepping Stones and Creating Futures Plus: A pilot randomised controlled trial of a co-developed intervention with young South Africans. PLOS Glob Public Health. 2025 Apr 23;5(4):e0004494. doi: 10.1371/journal.pgph.0004494. eCollection 2025. PMID 40267104